CLINICAL TRIAL: NCT05088200
Title: A Retrospective Case Series Study for Acute Abdomen in General Surgery Ward
Status: Completed | Type: Observational
Sponsor: Ahmadullah Danish (Other)
Responsible Party: Sponsor-Investigator, Ahmadullah Danish, A retrospective case series study for acute abdomen in general surgery ward of Aliabad teaching hospital, Kabul University of Medical Sciences
Organization: Kabul University of Medical Sciences (Other)
Other Study IDs: 118
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: The Study Was Aimed to Assessing the Clinical Profile of Acute Abdomen and Their Frequency According to Age and Sex
Keywords: Acute abdomen, Abdominal pain, Acute appendecitis, intestinal obstruction
MeSH Terms: conditions — Coitus; Abdomen, Acute; Abdominal Pain; Intestinal Obstruction | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — Our study is observational and we use secondary data

SUMMARY:
The acute abdomen is a clinical situation in which an acute an change in the condition of intra-abdominal organ, commonly attached to inflammation or infection need urgent and correct diagnosis .

DETAILED DESCRIPTION:
A special data collection sheet designed to collect data regarding the diagnosis, age and sex from the profile of patients retrospectively. Data entry was performed by using Microsoft Excel and all the data were analysed by SPSS.

ELIGIBILITY:
Inclusion Criteria:

* All of patients with acute abdomen that is admitted in general surgery ward of Aliabad teaching hospital.

Exclusion Criteria:

* traumatic abdominal injury, abdominal pain due to urological and gynaecological origin.

Ages: 15 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of patients with acute abdomen that is admitted in general surgery ward of Aliabad.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
A retrospective case series study for acute abdomen in general surgery ward of Aliabad teaching hospital | 21 March 2018-21 March 2019

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmadullah Danish, Kabul, Afghanistan

IPD SHARING:
Plan to Share IPD: Yes